CLINICAL TRIAL: NCT02936180
Title: Improving Influenza Immunization Responses in Rheumatoid Arthritis: A Strategy To Enhance Protection Against A Preventable Cause Of Death In An At Risk Population?
Brief Title: Standard Versus High Dose Inactivated Influenza Vaccine in RA
Acronym: IV-RA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: The Arthritis Society, Canada (Other)
Responsible Party: Principal Investigator, Ines Colmegna, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MP-37-2017-2773
Record Dates: First submitted 2016-10-07; First posted 2016-10-18 (Estimated); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Flu vaccine; Influenza
MeSH Terms: conditions — Arthritis, Rheumatoid; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard dose influenza vaccine (Active Comparator): Patients will receive one dose of FLUZONE® Standard Dose Quadrivalent Inactivated Influenza Vaccine (SD-QIV)
  Interventions: Biological: SD-QIV
- High dose influenza vaccine (Active Comparator): Patients will receive one dose of FLUZONE® High Dose Trivalent Inactivated Influenza Vaccine (HD-TIV)
  Interventions: Biological: HD-TIV

INTERVENTIONS:
Biological: HD-TIV
  Arms: High dose influenza vaccine
Biological: SD-QIV
  Arms: Standard dose influenza vaccine

SUMMARY:
Patients with rheumatoid arthritis have increased risk of seasonal influenza and influenza-related complications but have reduced vaccine immunogenicity. It is unknown whether patients with rheumatoid arthritis would benefit from more immunogenic vaccine formulations. This study investigated the immunogenicity and safety of a high-dose trivalent inactivated influenza vaccine (HD-TIV) in patients with rheumatoid arthritis compared to a standard-dose quadrivalent influenza vaccine (SD-QIV).

DETAILED DESCRIPTION:
Influenza, a vaccine-preventable respiratory disease, is ranked 8th among the causes of death in the Canadian population. Among rheumatoid arthritis (RA) patients, the incidence of both seasonal influenza and serious influenza-related illness (IRI) are increased. Despite being a high priority group targeted for vaccination, the diagnosis of RA and other patient-specific factors (i.e. older age, treatment, current smoking) are linked to impaired vaccination responses.

Thus the burden of influenza among people with RA is disproportionally high, and interventions to improve responses to influenza vaccination are urgently needed. Strategies to optimize protection in another vulnerable group, the elderly, include the use of quadrivalent vaccines, higher antigen doses, and adjuvants. A high-dose, trivalent, inactivated influenza vaccine (HD-TIV) has recently been shown to have a similar safety profile to standard dose vaccine (SD-TIV) with improved immunogenicity and protection in adults ≥65 years of age. Whether or not analogous strategies to improve responses to influenza vaccine will enhance protection in people with RA is unknown. The investigators hypothesize that the use of the HD-influenza vaccine will improve vaccine-induced protection (i.e. seroconversion and seroprotection) in people with RA compared to SD-influenza vaccine. The investigators propose to conduct a stratified, randomized, modified double blind, active-controlled trial to assess immune responses to two commercial influenza vaccines containing different antigen doses in individuals with RA.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of seropositive RA (rheumatoid factor (RF) and/or anti-CCP antibody positive) based on the 2010 ACR-EULAR criteria.
2. At least 6 months of treatment including anti-TNF agents, abatacept, rituximab (dose received within the previous 6 months) and/or methotrexate.
3. Informed consent form signed and dated.
4. Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

1. Vaccination against influenza in the 6 months preceding the trial vaccination.
2. Systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to TIV or to a vaccine containing any of the same substances.
3. History of Guillain-Barré syndrome within six weeks of a previous influenza vaccination.
4. Dementia or any other cognitive condition that could interfere with the trial procedures.
5. Thrombocytopenia or bleeding disorder contraindicating IM vaccination (according to treating rheumatologist).
6. Current alcohol abuse or drug addiction.
7. Moderate or severe acute illness with or without fever. If this exists, vaccination will be deferred until the individual has been medically stable and/or afebrile for at least 24 hours.
8. Signs and symptoms of an acute infectious respiratory illness. If this exists, vaccination will be deferred until the symptoms resolve.
9. Pregnant women (the rationale for excluding this group is not their lack of indication for vaccination but the changes of maternal immune responses during pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2016-10; Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ines Colmegna, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Colmegna I, Useche ML, Rodriguez K, McCormack D, Alfonso G, Patel A, Ramanakumar AV, Rahme E, Bernatsky S, Hudson M, Ward BJ. Immunogenicity and safety of high-dose versus standard-dose inactivated influenza vaccine in rheumatoid arthritis patients: a randomised, double-blind, active-comparator trial. Lancet Rheumatol. 2020 Jan;2(1):e14-e23. doi: 10.1016/S2665-9913(19)30094-3. Epub 2019 Nov 20. PMID 38258270
- See also: Publication — https://doi.org/10.1016/S2665-9913(19)30094-3

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Dose Influenza Vaccine: Patients will receive one dose of FLUZONE® Standard Dose Quadrivalent Inactivated Influenza Vaccine (SD-QIV)
  SD-QIV
- High Dose Influenza Vaccine: Patients will receive one dose of FLUZONE® High Dose Trivalent Inactivated Influenza Vaccine (HD-TIV)
  HD-TIV
Period: Overall Study
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Started | 140 | 139
Completed | 127 | 121
Not Completed | 13 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine | Total
Number analyzed (Participants) | 136 | 138 | 274
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 85 | 162
  >=65 years | 59 | 53 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (11.8) | 59.7 (13.9) | 60.8 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 109 | 218
  Male | 27 | 29 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 13 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 106 | 110 | 216
  More than one race | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Rate to HD- Versus SD-IV in People With RA
Description: Seroconversion rate (SCR): proportion of subjects in a given treatment group (SD- or HD) with either a ≥4-fold increase in reciprocal HI titres between D0 and D28 or a rise of undetectable HI titre (i.e. <1:10) pre-vaccination (D0) to an HI titre of ≥1:40 at D28 post vaccination.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Number analyzed (Participants) | 136 | 138
Participants | 12 | 31

2. Primary Outcome: Seroprotection Rate to HD- Versus SD-IV in People With RA
Description: Seroprotection rate (SPR): the proportion of subjects in a given treatment group attaining a reciprocal HI titre of ≥1:40 at D28 post-vaccination.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Number analyzed (Participants) | 136 | 138
Participants | 42 | 67

3. Primary Outcome: Geometric Mean Titres (GMTs) of HI in People With RA Who Received HD- Versus SD-IV
Description: Geometric mean titres (GMTs) of HI at D28.
Time Frame: Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Number analyzed (Participants) | 136 | 138
titer | 1.56 [1.22 to 1.90] | 2.06 [1.12 to 3.00]

4. Secondary Outcome: Durability of Detectable Levels of HI Antibody for SD- and HD- IV.
Description: Number of participants with detectable HI antibodies at Day 186
Time Frame: Day 186
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Number analyzed (Participants) | 127 | 121
Participants | 29 | 43

5. Secondary Outcome: Rates of Side Effects During the Surveillance Period in SD- and HD-IV.
Description: Number of Participants with Side Effects
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
Number analyzed (Participants) | 136 | 138
Participants | 19 | 20

6. Other Pre Specified Outcome: Performance of the Micro-neutralization Assay in Comparison to the HI Assay.
Time Frame: Day 186
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Rates of Health Care Use in Patients Receiving SD- or HD-IV.
Time Frame: Day 186
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Standard Dose Influenza Vaccine | High Dose Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 1/136 | 2/138
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/138
Other Adverse Events (participants affected / at risk) | 14/136 | 19/138
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dose Influenza Vaccine (N=136) | High Dose Influenza Vaccine (N=138)
Unsolicited adverse events (Respiratory, thoracic and mediastinal disorders) | 14 | 19 — Respiratory illness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT02936180/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT02936180/SAP_001.pdf